CLINICAL TRIAL: NCT06330285
Title: Comparison of E-Learning and Face-to-Face Learning in Cardiopulmonary Exercise Test Training: Randomized Controlled Study
Brief Title: Comparison of E-Learning and Face-to-Face Learning in Cardiopulmonary Exercise Test Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Havva Talay Çalış, Professor Doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: e learning pgme/cpet
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Exercise Test; Learning
Keywords: E-Learning; Face-to-Face Learning; Cardiopulmonary Exercise Test Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): e-learning
  Interventions: Other: e-learning
- Group 2 (Active Comparator): face to face learning
  Interventions: Other: face to face learning

INTERVENTIONS:
Other: e-learning — CPET (Cardiopulmonary exercise test) e-learning application The content, planning and design of 4 lessons are as follows:
  1. Introduction and CPET Fundamentals:
  2. Respiratory function tests
  3. Field Field Tests and CPET Results
  4. Problems and examples
  Other Names: e- education
  Arms: Group 1
Other: face to face learning — CPET (Cardiopulmonary exercise test) face to face education. The content, planning and design of 4 lessons are as follows:
  Contents:
  1. Introduction and CPET Fundamentals:
  2. Respiratory function tests
  3. Field Field Tests and CPET Results
  4. Problems and examples
  Other Names: face to face education
  Arms: Group 2

SUMMARY:
The main purpose of this study is to compare the effect of teaching Cardiopulmonary Exercise Test (CPET) via e-learning and face-to-face to doctors receiving postgraduate medical education (PGME).

DETAILED DESCRIPTION:
CPET is the most objective and valuable test for the cardiopulmonary rehabilitation (CPR) program to be planned for back-up for patients with cardiopulmonary diseases.

CPET is performed in a small number of centers in Turkey, in Physical Medicine and Rehabilitation (PTR) Units. Depending on the equipment available during specialty training, not all specialty students can access this training.

CPET is the first test performed for planning cardiopulmonary rehabilitation (CPR). According to the results, an appropriate CPR plan is made for the patient.

CPET indications, contraindications, application of the test, evaluation of the test with patient samples, and appropriate interventions for complications that may develop during the test are important.

It is important that all specialist students have access to this training. The aim of this study is; To evaluate the impact of e-learning with PGME and to reach all specialist students in the future, if necessary, based on the results.

The focus of this study is to examine the changes in doctors' success levels, motivations, distance education attitudes, cognitive flexibility and anxiety levels, especially in the pre- and post-training periods, and to compare these changes with face-to-face training.

ELIGIBILITY:
Inclusion Criteria:

* Those who gave consent,
* Graduates of the Faculty of Medicine and currently receiving specialist training,
* Those who can do what the training requires during the training period (participating in live classes, answering scales, etc.)

Exclusion Criteria:

* Those who cannot attend the training program regularly
* In addition, those who cannot attend more than 4 classes with or without an excuse will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-22 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Open-Ended Achievement Test | at baseline, After the training is completed (at the 4. week)
  Open-Ended Achievement Test: It is used to measure doctors' knowledge and skill levels on CPET. It will be prepared by the trainers for each lesson.
Adult Motivation Scale | at baseline, After the training is completed (at the 4. week)
  Used to evaluate doctors' motivation towards the training process. The purpose of the scale is to determine the motivation levels and orientations of adults. It consists of two factors and 21 items in total. In the analyzes conducted for the reliability of the scale, the Cronbach Alpha reliability coefficient was found to be 0.94. This value shows that the scale has high internal consistency.
Distance Education Attitude Scale in Lifelong Learning | at baseline, After the training is completed (at the 4. week)
  It is used to measure doctors' attitudes towards distance education. "Distance Education Attitude Scale in Lifelong Learning" is designed to evaluate attitudes towards distance education.
Cognitive Flexibility Scale | at baseline, After the training is completed (at the 4. week)
  Used to evaluate doctors' ability to solve problems, adapt and respond to different situations. The Cognitive Flexibility Scale (CFS) is used to measure how individuals adapt their behavior to new and unexpected situations occurring in their environment. CFS was developed by Dennis and Vander Wall and adapted into Turkish. CFs is a self-report type assessment tool with a total of 20 items, consisting of 'alternatives' and 'control' subscales. Cronbach's alpha value of the Alternatives subscale at the first and last measurement was .91. Cronbach's alpha values of the control subscale are .86 in the first measurement and .84 in the last measurement.
State and Trait Anxiety Scale | at baseline, After the training is completed (at the 4. week)
  It is used to measure the momentary and continuous anxiety states of doctors during the training process. This scale is used to evaluate individuals' momentary and persistent anxiety states. State Anxiety and Trait Anxiety. There are 20 items in the state anxiety scale. There are 20 more items in the trait anxiety scale. There are 40 items in the scale in total. Kuder-Richardson reliability of the inventory was .83 to .87 for the Trait Anxiety Subscale; For the State Anxiety Subscale, it was found to be between .94 and .96. Item reliability correlations were .34 to .72 for the Trait Anxiety Subscale; For the State Anxiety Subscale, the range between .42 and .85 indicates that the Turkish translated items are reliable. The test-retest reliability rates of the inventory are .71 to .86 for the Trait Anxiety Subscale; For the State Anxiety Subscale, it is between .26 and .68 and is considered sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: HAVVA TALAY ÇALIŞ, Study Director — Health Sciences University, Kayseri Medical Faculty

IPD SHARING:
Plan to Share IPD: No